CLINICAL TRIAL: NCT01573546
Title: Lifestyle, CVD Risk, and Cognitive Impairment
Brief Title: ENLIGHTEN: Exercise and NutritionaL Interventions for coGnitive and Cardiovascular HealTh ENhancement
Acronym: ENLIGHTEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00031464
Record Dates: First submitted 2011-12-22; First posted 2012-04-09 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Cognitive Impairment, no Dementia (CIND)
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise; Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Aerobic Exercise (Experimental)
  Interventions: Behavioral: Aerobic Exercise
- DASH diet (Experimental)
  Interventions: Behavioral: DASH diet
- Combined aerobic exercise and DASH diet (Experimental)
  Interventions: Behavioral: Aerobic Exercise; Behavioral: DASH diet
- Health education control (Active Comparator)
  Interventions: Other: Health education control

INTERVENTIONS:
Behavioral: Aerobic Exercise — Participants will exercise for 6 months. In the initial 3-month supervised phase, patients will exercise 3 times a week at a level of 50-75% of their initial peak heart rate reserve (HRR) or at their peak heart rate without symptoms, or ST-segment depression > 1 mm, as determined at the time of their initial exercise test. Aerobic exercise consists of 10 minutes of warm-up exercises followed by 30 minutes of continuous walking or (stationary) biking. Each exercise session will conclude with a 10 minute period of cool-down exercises. During weeks 13 to 24 (i.e., home maintenance phase), participants will be asked to perform 3 aerobic sessions per week at home at 60-70% HRR.
  Arms: Aerobic Exercise; Combined aerobic exercise and DASH diet
Behavioral: DASH diet — Participants in the DASH condition only receive instruction in modifying the content of their diet to meet DASH guidelines. Participants will be explicitly asked not to exercise and to focus their attention on what they eat. Participants will have been told (in the initial consent form) that the study is designed to study effects of two interventions (altering diet content and exercise) both of which have been shown to improve health. Participants will also be told that it may be easier or more effective for them if they focus first on learning to alter diet content, and they are free to exercise at the end of the 6-month period. Following an initial 1-day feeding period, participants, along with their study partners, will receive instruction on the DASH diet and feedback on their adherence to the diet in a series of half-hour, weekly small group sessions (3 to 4 participants).
  Arms: Combined aerobic exercise and DASH diet; DASH diet
Other: Health education control — The Health Education control group will receive weekly 30-min lectures on relevant, health-related topics but will not receive instruction in the DASH diet nor will exercise be promoted. These participants will be asked to maintain their usual dietary and exercise habits for 6 months until they are re-evaluated. These sessions are designed to provide useful information about medical aspects of CVD, but will not provide instruction in the DASH diet or exercise.
  Arms: Health education control

SUMMARY:
ENLIGHTEN will examine the effects of exercise, the dietary approaches to stop hypertension diet (DASH), and a combined exercise and DASH intervention on cognitive function among adults with cardiovascular disease (CVD) risk and cognitive deficits. Participants will be randomized to one of the three treatments, or a health education control condition, for 6 months, and will complete assessments of CVD health and cognitive function before and after treatment.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death and disability in the United States, affecting more than 81 million American adults. It is well established that risk factors such as hypertension, diabetes, and hyperlipidemia not only place individuals at risk for CVD, but also place them at risk for neurocognitive impairment and dementia. CVD risk factors have been shown to be associated with a cascade of neurophysiologic and neuroanatomic changes, resulting in cognitive impairment and dementia. Exercise and diet have been shown to improve CVD risk factors and also appear particularly promising lifestyle approaches for preventing dementia among individuals at risk, such as those with cognitive impairment, no dementia (CIND). ENLIGHTEN is a randomized clinical trial of diet and exercise among patients with CIND.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years or older
* Sedentary
* Score of 19-25 on the Montreal Cognitive Assessment Battery or verbal fluency score of =< 12 or animal fluency score of =<15
* At least one cardiovascular risk factor (hypertension, diabetes, cholesterol, obesity, current smoking, or family history) or a documented history of cardiac disease (myocardial infarction, coronary artery bypass grafting, peripheral vascular disease, >70% stenosis, or mild stroke without residual deficit)

Exclusion Criteria:

* Any significant neurological disease other than CIND, such as Parkinson's disease, multi-infarct dementia, Huntington' s disease, progressive supranuclear palsy, brain tumor, normal pressure hydrocephalus, subdural hematoma, seizure disorder, multiple sclerosis, or history of head trauma with persistent neurological deficits
* Psychotic disorder within the past two years (DSM IV criteria) or acutely suicidal
* History of alcohol or substance abuse or dependence within the past two years (DSM IV criteria)
* History of schizophrenia
* Any significant systemic illness or unstable medical condition that could lead to difficulty in complying with the protocol including a history of systemic cancer within the past 5 years (nonmetastatic skin cancers are acceptable)
* Myocardial infarction (within the past 3 months) or unstable or severe congestive heart failure (e.g. class III-IV heart failure)
* End-stage pulmonary disease; uncontrolled diabetes mellitus or uncontrolled hypertension(systolic BP>170 or diastolic BP >100 mm Hg on medication)
* Musculoskeletal disorders precluding the ability to exercise (e.g. severe arthritis)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-12; Primary Completion 2016-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in Executive Function | Baseline to post-treatment assessment at 6 months
  Composite executive function measure includes Trail Making Test, Stroop Test, Digit Span, Digit Symbol Substitution Test, Ruff 2 & 7 Test, and Animal Naming Test

SECONDARY OUTCOMES:
Change in Memory | 6 months
  Secondary outcomes will include composite measures of memory (Hopkins Verbal Learning Test-Revised and Medical College of Georgia Complex Figure Test)
Change in Language | 6 months
  Secondary outcomes will include composite measures of language (Controlled Oral Word Association Test and Animal Naming Test)
Inflammation | 6 months
  We will also assess treatment effects on measures of inflammation, including C-reactive protein and interleukin-6.
Functional Capacity | 6 months
  Functional capacity (6MWT and peak VO2). Six-minute walk distance (6MWT) and peak VO2 from a treadmill test will be assessed by an exercise physiologist.
Blood Pressure | 6 months
  We also will examine treatment effects on the vascular function measures, including blood pressure.
Flow-mediated dilation of the brachial artery | 6 months
  We also will examine treatment effects on the vascular function measures, including flow-mediated dilation of the brachial artery.
Arterial Stiffness | 6 months
  We also will examine treatment effects on the vascular function measures, including pulse-wave velocity of the femoral artery.
Intima-medial thickness | 6 months
  We also will examine treatment effects on the vascular function measures, including intima-medial thickness of the carotid artery.
Fasting glucose | 6 months
  We will also assess treatment effects on measures fasting glucose
Cholesterol | 6 months
  We will also examine treatment effects on cholesterol, including LDL, HDL, and total cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: James A Blumenthal, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Blumenthal JA, Smith PJ, Welsh-Bohmer K, Babyak MA, Browndyke J, Lin PH, Doraiswamy PM, Burke J, Kraus W, Hinderliter A, Sherwood A. Can lifestyle modification improve neurocognition? Rationale and design of the ENLIGHTEN clinical trial. Contemp Clin Trials. 2013 Jan;34(1):60-9. doi: 10.1016/j.cct.2012.09.004. Epub 2012 Sep 19. PMID 23000080
- [Derived] Blumenthal JA, Smith PJ, Mabe S, Hinderliter A, Welsh-Bohmer K, Browndyke JN, Doraiswamy PM, Lin PH, Kraus WE, Burke JR, Sherwood A. Longer Term Effects of Diet and Exercise on Neurocognition: 1-Year Follow-up of the ENLIGHTEN Trial. J Am Geriatr Soc. 2020 Mar;68(3):559-568. doi: 10.1111/jgs.16252. Epub 2019 Nov 22. PMID 31755550
- [Derived] Blumenthal JA, Smith PJ, Mabe S, Hinderliter A, Lin PH, Liao L, Welsh-Bohmer KA, Browndyke JN, Kraus WE, Doraiswamy PM, Burke JR, Sherwood A. Lifestyle and neurocognition in older adults with cognitive impairments: A randomized trial. Neurology. 2019 Jan 15;92(3):e212-e223. doi: 10.1212/WNL.0000000000006784. Epub 2018 Dec 19. PMID 30568005
- [Derived] Blumenthal JA, Smith PJ, Mabe S, Hinderliter A, Welsh-Bohmer K, Browndyke JN, Lin PH, Kraus W, Doraiswamy PM, Burke J, Sherwood A. Lifestyle and Neurocognition in Older Adults With Cardiovascular Risk Factors and Cognitive Impairment. Psychosom Med. 2017 Jul/Aug;79(6):719-727. doi: 10.1097/PSY.0000000000000474. PMID 28437380